CLINICAL TRIAL: NCT02107989
Title: Noninvasive Pre-surgical Evaluation of Patients With Focal Epilepsy and Establishment of a Normative Imaging Database
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140061; 14-N-0061
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-09-25

CONDITIONS: Epilepsy
Keywords: Epilepsy; MRI; fMRI; MEG; Natural History
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: healthy volunteers
  Interventions: Device: MRI; Device: MEG
- Patients: Patients
  Interventions: Device: MRI; Device: MEG

INTERVENTIONS:
Device: MRI — MRI of the brain is routinely used to identify abnormal areas of cortex in patients with medically refractory epilepsy. MRI evaluations of brain may be performed at field strengths of 1.5T, 3T, and/or 7T, under conditions designated by the FDA as constituting nonsignificant risk.
Device: MEG — MEG/EEG: Magnetoencephalography (MEG) is commonly used during epilepsy pre-surgical evaluations to help with localizing epileptic foci. MEG will be obtained as clinically indicated, usually in patients with unclear seizure focus localization who are undergoing presurgical evaluation, particularly when they have frequent interictal discharges on EEG. MEG records very small magnetic fields generated by the brain at rest, or in response to a task or to epileptic activity. Resting state MEG/EEG analysis will be used for research purposes only.

SUMMARY:
Objectives:

The overall study objective is to compare the sensitivities and specificities of morphometric analysis techniques using structural MRI images based on pre- and postsurgical localization of epileptic foci in patients undergoing presurgical evaluation for medically refractory epilepsy. To carry out these analyses, we aim to establish an age-stratified normative imaging database using healthy volunteers. Additional objectives are to identify abnormal networks in these patients using resting state fMRI/EEG and MEG/EEG, and to use language and memory fMRI tasks to examine the effects of epileptogenic zones and surgery on cognitive function and the networks associated with these functions.

Study population:

300 adults and children (age 8 and older) with uncontrolled focal epilepsy, and 200 age-stratified healthy volunteers.

Design: A retrospective and prospective natural history study. Research procedures for patients in this study include neuropsychological testing and 1-4 MRI sessions during presurgical evaluation and an additional 1-3 MRI sessions and neuropsychological testing approximately 12 months post-operatively. Research testing (such as research neuropsychological tests or MRI scanning sequences) will be done during a visit for clinical testing whenever possible, likely reducing the number of required visits. Patients will also have optional MEG and 7T structural imaging. Data will also be obtained from patients who have already undergone epilepsy surgery if they had procedures as outlined in the protocol and are willing to share the data. Healthy volunteers will receive a subset of the pre-operative procedures for patients, requiring at least 3 visits. In order to ensure adequate data acquisition, subjects may be re-scanned up to three times for the portions of the study in which they participated, possibly requiring additional visits.

Outcome measures:

The main outcomes will be establishment of normative values for morphometric analysis methods in age-stratified normal controls, and comparison of the sensitivity and specificity of these measures to pre- and postsurgical localization of the epileptogenic zone. Secondary outcome measures will include determination of the sensitivity and specificity of source localization using MEG/EEG and resting state fMRI/EEG, and to evaluate changes in activation during rest, as well as language and memory fMRI tasks in patients pre- and postsurgically, to examine the effects of epileptogenic zones and surgery on cognitive function and the networks underlying these functions.

...

DETAILED DESCRIPTION:
Objectives: The overall study objectives of this study are 1) to establish an age-stratified normative imaging database, 2) to explore the use of non-invasive imaging techniques such as morphometric analysis of structural MRI, resting state fMRI/EEG and resting state MEG/EEG to localize seizure foci. The sensitivities and specificities of analysis techniques will be determined based on pre- and postsurgical localization of epileptic foci in patients undergoing presurgical evaluation for medically refractory epilepsy. Additional objectives are to identify abnormal networks in these patients using resting state fMRI/EEG and MEG/EEG, to explore the use of language and memory fMRI tasks to examine the effects of epileptogenic zones and surgery on cognitive function and the networks associated with these functions, and to explore whether changes in resting state and task-based fMRI networks can be identified following epilepsy surgery, and how these changes relate to seizure and neuropsychological outcomes.

Study population: 500 adults and children (age 8 and up) with uncontrolled focal epilepsy, and 200 age-stratified healthy volunteers.

Design: A retrospective and prospective natural history study. Research procedures for patients in this study include 1-4 MRI sessions during presurgical evaluation and additional 1-3 MRI sessions approximately 12 months post-operatively. Research testing (such as research neuropsychological tests or MRI scanning sequences) will be done during a visit for clinical testing whenever possible, likely reducing the number of required visits. Patients will also have optional MEG, neuropsychological testing, fMRI and 7T structural imaging. Data will also be obtained from patients who have already undergone epilepsy surgery if they had procedures as outlined in the protocol and are willing to share the data. Healthy volunteers will receive a subset of the pre-operative procedures for patients, requiring at least 3 visits. In order to ensure adequate data acquisition, subjects may be re-scanned up to three times for the portions of the study in which they participated, possibly requiring additional visits.

Outcome measures:

The main outcomes will be establishment of normative values for morphometric analysis methods in age-stratified normal controls, with exploratory outcome measures of determination of comparison of the sensitivity and specificity of these measures to pre and postsurgical localization of the epileptogenic zone. Exploratory outcome measures include determination of the sensitivity and specificity of source localization using morphometric analysis of structural MRI, resting state MEG/EEG and resting state fMRI/EEG, evaluation of changes in activation during rest, as well as language and memory fMRI tasks in patients pre- and post-surgically, and examination of the effects of epileptogenic activity and surgery on cognitive function and the networks underlying these functions.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PATIENTS:
* Age 8 and older
* Evaluated or under evaluation for epilepsy surgery under protocol 18-N-0066,11-N-0051 or 16-N-0041
* Documentation of focal epilepsy based on MRI, EEG and/or ictal semiology
* Ability to give informed consent, have or be able to assign a legally authorized representative able to give consent (for adults without consent capacity), or parent/guardian able to provide informed consent (for a child).

INCLUSION CRITERIA FOR PATIENTS SOLELY CONTRIBUTING DATA:

* Had epilepsy surgery with presurgical evaluation under 18-N-0066
* Age 8 and up at the time of epilepsy surgery evaluation
* Had a preoperative structural brain MRI of the type used in this protocol

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Age 8 and older
* Ability to give informed consent or have a parent/guardian able to provide informed consent if a child.
* Ability to cooperate with MRI scanning without anesthesia

EXCLUSION CRITERIA FOR PATIENTS:

* Contraindications to MRI or MEG studies (such as pacemakers, cochlear implants, shrapnel, permanent eyeliner)
* Claustrophobia or anxiety disorders exacerbated by the MRI scanner
* Pregnancy. All females of childbearing potential must have a negative pregnancy test prior to MRI scanning

EXCLUSION CRITERIA FOR PATIENTS SOLELY CONTRIBUTING DATA:

-Not able or willing to give consent or do not have an appropriate surrogate who can provide consent

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Contraindications to MRI or MEG studies (such as pacemakers, cochlear implants, shrapnel, permanent eyeliner)
* Claustrophobia or anxiety disorders exacerbated by the MRI scanner
* Significant medical conditions that may affect the central nervous system, such as psychiatric disorders (such as mood disorders, psychotic disorders, substance abuse or dependence), significant neurologic disorders (such as brain injury, neurodegenerative disorders, multiple sclerosis, stroke, movement disorders, epilepsy), or active systemic disease that may affect the central nervous system (such as uncontrolled hypertension, autoimmune disorders or other inflammatory disorders, neoplastic disease)
* Use of centrally acting medications in the past 6 weeks, such as benzodiazepines, barbiturates, antidepressants, beta-blockers, and drugs for treating epilepsy or migraine
* Pregnancy. All females of childbearing potential must have a negative pregnancy test prior to MRI scanning

Ages: 8 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 500 adults and children (age 8 and up) with uncontrolled focal epilepsy, and 200 age-stratified healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2014-03-11 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
All outcomes in this study are Exploratory. | All outcomes in this study are Exploratory.
  All outcomes in this study are Exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Inati, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-N-0061.html